CLINICAL TRIAL: NCT05679245
Title: Prevalence of Post-traumatic Stress Disorder and Trauma-related Symptoms in a Sample of Healthy Controls in the Barcelona Region of Catalonia, Spain
Brief Title: Prevalence of Post-traumatic Stress Disorder and Trauma Symptoms in a General Population Sample
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Other Study IDs: CS01
Record Dates: First submitted 2022-12-21; First posted 2023-01-10 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2022-12

CONDITIONS: Post-traumatic Stress Disorder; Psychological Trauma
Keywords: post-traumatic stress disorder; psychological trauma; healthy controls
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Psychological Trauma | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Controls: Healthy controls without mental disorder in the general population of the Barcelona area of Catalonia, Spain to be assessed for exposure to traumatic life events, post-traumatic stress disorder, trauma symptoms, dissociative symptoms, affective symptoms, and psychosocial functioning.
  Interventions: Diagnostic Test: Assessment for exposure to psychological trauma and related symptoms

INTERVENTIONS:
Diagnostic Test: Assessment for exposure to psychological trauma and related symptoms — To be assessed for exposure to traumatic life events, post-traumatic stress disorder, trauma-related symptoms, dissociative symptoms, affective symptoms, and psychosocial functioning.

SUMMARY:
The goal of this observational study is to learn about how many people have post-traumatic stress disorder and related symptoms in the general population of people without any mental illness in the Barcelona region of Catalonia, Spain. The main questions it aims to answer are:

* What is the prevalence of post-traumatic stress disorder in a sample of healthy controls without other mental disorders?
* What is the prevalence of trauma-related symptoms in a sample of healthy controls without mental illness?
* What is the prevalence of dissociative symptoms (including symptoms of depersonalisation and somatoform dissociation) in a sample of healthy controls without mental illness?
* What is the prevalence of recent and childhood traumatic life events in a sample of healthy controls without mental illness?
* What is the prevalence of difficulties in psychosocial functioning in healthy controls without mental illness?
* What is the prevalence of depressive symptoms in healthy controls without mental illness?
* What is the prevalence of general psychiatric symptoms in healthy controls without mental illness? Participants will be asked to take part in an online screening programme, and then to come to an interview with a clinician who will apply validated scales to test the above.

DETAILED DESCRIPTION:
This is a study to provide normative data for the prevalence of traumatic life events, post-traumatic stress disorder and trauma-related symptoms, and their impact on psychosocial functioning, and affective symptoms in healthy controls (i.e. without mental illness) in the Barcelona region of Catalonia, Spain.

ELIGIBILITY:
Inclusion Criteria:

* to be an adult (18-65 years inclusive)

Exclusion Criteria:

* to have a mental disorder except for post-traumatic stress disorder, determined by application of the Mini International Neuropsychiatric Interview (MINI)
* active suicidal ideation
* presence of organic brain disease
* presence of somatic diseases such as fibromyalgia or chronic fatigue syndrome
* presence of autoimmune diseases such as HIV or AIDS

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult controls without mental disorder from the Barcelona region of Catalonia, Spain.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Prevalence of post-traumatic stress disorder in a sample of healthy controls without mental disorder | cross-sectional, baseline
  Prevalence of post-traumatic stress disorder according to criteria of the Diagnostic and Statistical Manual of Mental Disorders - 5th Edition, as per the Global Evaluation of Post-traumatic Stress Disorder Scale (EGEP-5), which assesses the presence or absence of post-traumatic stress disorder.
Prevalence of trauma symptoms in a sample of healthy controls without mental disorder | cross-sectional, baseline
  Prevalence of trauma-related symptoms according to the Impact of Events Scale-Revised (IES-R), which is scored on a Likert scale with a maximum score of 110, with higher scores meaning a greater level of trauma symptoms.
Prevalence of dissociative symptoms in a sample of healthy controls without mental disorder | cross-sectional, baseline
  Prevalence of dissociative symptoms according to the Dissociative Experiences Scale (DES). The final score is out of 100, with higher scores meaning a greater number of symptoms.

SECONDARY OUTCOMES:
Prevalence of depressive symptoms in a sample of healthy controls without mental disorder | cross-sectional, baseline
  Prevalence of depressive symptoms according to the Hamilton Depression Rating Scale (HDRS), which can provide a total score between 0 and 63, with higher scores meaning greater depressive symptoms.
Prevalence of psychiatric symptoms in a sample of healthy controls without mental disorder | cross-sectional, baseline
  Prevalence of psychiatric symptoms according to the Brief Psychiatric Rating Scale (BPRS). The first 18 items on this scale provide a total score from 0 to 146, with higher scores signifying more severe psychiatric symptoms, while item 19 provides an estimate of severity of illness on a Likert scale from 1 to 7.
Prevalence of symptoms of somatoform dissociation in a sample of healthy controls without mental disorder | cross-sectional, baseline
  Prevalence of symptoms of somatoform dissociation according to the Somatoform Dissociation Questionnaire (SDQ-20). Each item is scored on a Likert scale from 1 to 5, up to a total score of 100. Higher scores denote more somatoform symptoms.
Prevalence of depersonalisation dissociative symptoms in a sample of healthy controls without mental disorder | cross-sectional, baseline
  Prevalence of depersonalisation dissociative symptoms according to the Cambridge Depersonalisation Scale. Each item is scored for frequency (0 to 4) and duration (1 to 6), and these scores are summed together to create a total score. Higher scores indicate greater levels of dissociative symptoms.
Prevalence of difficulties in psychosocial functioning in a sample of healthy controls without mental disorder | cross-sectional, baseline
  Prevalence of difficulties in psychosocial functioning according to the Functioning Assessment Short Test (FAST). Each item on this scale is scored on a Likert scale of 0 to 3, providing a total score between 0 and 72. Higher scores indicate a greater degree of difficulty in functioning.
Prevalence of childhood trauma events (physical, sexual, or emotional abuse, and physical or emotional neglect) in a sample of healthy controls without mental disorder | cross-sectional, baseline
  Prevalence of childhood trauma experiences according to the Childhood Trauma Questionnaire (CTQ). This scale provides a score for each subscale of physical, sexual, or emotional abuse, and physical or emotional neglect, with scores categorised as ranging from none to severe.
Prevalence of recent stressful life events in a sample of healthy controls without mental disorder | cross-sectional, baseline
  Prevalence of recent stressful life events in the previous year according to the Social Readjustment Rating Scale (Holmes & Rahe). This scale provides the number of stressful events. Each event has a weighted score which is summed to create a total score, with higher scores signifying a greater risk of stress-related illness.

CONTACTS AND LOCATIONS:
Locations (1):
- Alicia Valiente, Barcelona, Spain